CLINICAL TRIAL: NCT04099615
Title: New Predictive Biomarkers of Functional Recovery Prior the Endovascular Treatment of Acute Ischemic Stroke. PROMISE (Somatosensory Evoked POtEntials MonItoring During Acute Ischemic StrokE) Study
Brief Title: PROMISE (Somatosensory Evoked POtEntials MonItoring During Acute Ischemic StrokE) Study
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Sponsor
Other Study IDs: 201708.10
Record Dates: First submitted 2019-08-17; First posted 2019-09-23 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Acute Cerebrovascular Accident; Endovascular Procedures
Keywords: Evoked Potentials, Somatosensory; Acute Cerebrovascular Accident; Endovascular Procedures
MeSH Terms: conditions — Stroke | interventions — Evoked Potentials, Somatosensory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endovascular urgent stroke treatment group: Patients between 18 and 85 years old who have and acute cerebral stroke due to a demonstrated occlusion in the anterior circulation (M1 or M2 segment of middle cerebral artery with or without ipsilateral internal carotid artery (ICA), that undergo endovascular acute therapy fulfilling all inclusion criteria and with non exclusion criteria for that treatment. We also exclude patient with well-documented history of neuromuscular disorders, stroke or central nervous system tumors that could interfere in the SEPs assessment.
  Interventions: Procedure: Somatosensory Evoked Potentials

INTERVENTIONS:
Procedure: Somatosensory Evoked Potentials — We stimulate both median nerves at wrist by means of surface adhesive electrodes. We apply square wave electrical pulses of 0.2 ms duration at a frequency of 5.7Hz. SEPs are recorded in a referential fashion from the C3' and C4' positions and from a reference electrode at Fpz or Cz' electrodes(international 10-20 system) with needle electrodes. The target signal is the presence of N20 response ipsilateral to the stroke site and, if present, measure amplitude and latency comparing with the contralateral if present. SEPs are registered during the whole procedure.
  Other Names: SEP

SUMMARY:
Endovascular treatment in patients with acute ischemic stroke due to large vessel occlusion does not always lead to good clinical and functional outcome, despite achieving complete arterial recanalization. The rate of significant functional disability or death after three months of an acute ischemic stroke still ranges from 40% to 67%. There is experimental and clinical evidence that somatosensory evoked potentials (SEPs) are good indicators of cerebral blood flow.

The primary objective of this study is to determine the sensitivity and specificity of N20 response of SEPs prior to mechanical thrombectomy (MT) as a predictor of functional independence at 90 days after endovascular treatment. Secondly, the investigators will study whether SEPs may be neurophysiological markers of brain tissue in ischemic penumbra and optimal collateral circulation.

Bilateral median nerve SEPs will be recorded before and continuously during MT in patients with acute ischemic stroke and anterior large vessel occlusion. N20 response ipsilateral to the cerebral hemisphere affected will be measured (qualitatively and quantitatively). The adjusted predictive value of the N20 biomarker on functional independence after MT will be analyzed by binary logistic regression and its predictive value on the full range of disability by ordinal logistic regression. The investigators will construct different regression models with other clinical predictors available at the prehospital setting and with those determined after hospital admission to determine the independent predictive power of the N20 response for a potential treatment decision-making. Finally, the investigators will study whether SEP can be neurophysiological markers ischemic penumbra tissue and optimal collateral circulation through its correlation with multimodal neuroimaging techniques.

SEPs recording is non-invasive technique that can be performed at the bedside of the patient. The development of a portable device which could allow SEPs recording by sanitary staff (pre- and intrahospitally) would provide early data about N20 value, speeding up streamline decision making.

DETAILED DESCRIPTION:
PROMISE (somatosensory evoked PotEntials MonItoring during the acute ischemic StrokE) is a prospective, observational, single center study of somatosensory evoked potentials (SEPs) monitoring with blinded clinical and neuroimaging evaluation of a cohort of patients with acute ischemic stroke undergoing endovascular mechanical thrombectomy (MT). The study is conducted under clinical routine protocols following the ESO and ASA guidelines (29). All patients, or their surrogates, provide written informed consent for using their clinical data for the research purposes.

The study has been designed to confirm in a large cohort a diagnostic hypothesis previously tested in a pilot academic study. The invention, as a solution to a specific technological problem, novelty, usefulness, and non-obviousness, has been protected by an European patent. The pilot study was founded by our academic Institution. This confirmatory study aims to validate the presence of the N20 response on SEPs monitoring prior to- and during the mechanical thrombectomy (MT) as a non-invasive and useful biomarker of functional recovery after MT.

Patients Recruitment period has started in February 2018 and will be open until June 2020 since the project end is expected for December 2020. Eligible patients are older than 18 years with an score equal or less of 2 in the modified Rankin Scale, and an occlusion in the anterior circulation (M1 or M2 segment of middle cerebral artery with or without ipsilateral internal carotid artery (ICA) significant stenosis or occlusion diagnosed by CT angiography (CTA) or angio-MRI) The study site is a certified comprehensive stroke center (CSC) that treats more than 500 patients with acute stroke and performs more than 100 mechanical stroke thrombectomy procedures annually and is staffed by trained neurointerventional technique.

A sample of 228 patients has been estimated to be necessary to demonstrate the utility of SEPs. They are going to be recruited from acute stroke patients gone under urgent thrombectomy in our center. Data of the patient is going to be register manually on paper and electronically with a statistical program (SPSS).

Medical treatment and mechanical thrombectomy workflow. Intravenous alteplase is given within 4.5 hours in eligible patients following a model ship or drip and ship model with a DTN target median time of less than 35 min. The target time from hospital arrival at the CSC to groin puncture is 80 minutes or less and from study baseline neuroimaging to first reperfusion is 90 minutes or less. MT is performed with stent retrievers or thrombus aspiration. The use of general anesthesia or conscious sedation is left at the discretion of the neurointerventional staff, but conscious sedation is preferred over intubation (30,31). BP and vital signs are continuously monitored during the procedure. Patients are admitted at acute stroke units (or ICU if needed) and treated following the European Stroke Organization ESO guidelines(32)

Clinical and neuroimaging assessments All participants have standard assessments of demographic characteristics, medical history, laboratory values and stroke severity by means of NIHSS score at the moment of the admission. Time metrics from stroke onset to different diagnostic and treatment interventions will be recorded during the acute phase. Basal neuroimaging may be indistinctly noncontrast head computed tomography (NCCT) plus CTA, multiparametric MR or perfusion CT (CTP) if MR is not available. In patients whose vascular occlusion study confirming qualifying occlusion is performed beyond 4.5 hours of last seen well or when the neurointerventional team is not immediately available in-hospital, multiparametric MR or CTP are recommended prior to the endovascular treatment, although treatment decision is only made following the ASPECTS score criteria. Follow-up NCCT or MR scans are performed within 24 hours for assessment of infarct volume and to rule out intracranial hemorrhage or malignant edema. CTA, MRA or TCD are used to confirm persisting vessel revascularization at 24 hours.

CTP protocol is carried out on a 64 detector scanner (APV General Electrics, GE Medical Systems; Milwaukee, Wisconsin, USA) and includes CBF, CBV, MTT and TMax perfusion maps. MR protocol is carried out on a 3 Tesla Siemens Magneton Verio with a 32-Channel Head Coil. MR images include axial brain SWI/EPI-gradient recalled echo (GRE), DWI, fluid attenuation inversion recovery imaging (FLAIR), Angio MR TOF, dMRA (dynamic postcontrast MR angiography) and perfusion study, which is performed immediately after dynamic study. All images are anonymised and stored in DICOM format. Blinded investigators to clinical outcome and SEPs monitoring adjudicate all neuroimaging studies. Imaging investigators perform a visual analysis of qualitative variables and quantitative analysis of post-processed variables: firstpass permeability and perfusion maps. Post-process of DWI and perfusion sequences are done by using Olea Sphere platform. In addition, RAPID software (iSchemaView, Redwood City, CA) is used for emergent baseline and follow-up ischemic lesion volume calculation on MR-DWI or CTP-rCBF maps and for the automatic evaluation os ASPECTS score on NCCT and DWI-MR.

Pre-procedural imaging variables include volume and location of ischemic core and hypoperfused tissue at baseline, severity of hypoperfusion, site of occlusion and degree of collaterals according to the Arterial Collateral Grading Scale (ACG) if CTA or by using the ASITN/SIR Collateral Grading System scale if dMRA is performed. Follow-up images include volume and location of ischemic lesion, hemorrhagic transformation and arterial status.

Testing: SEPs monitoring Evoked potentials recordings are performed by the intraoperative monitoring system OSIRIS (Inomed Medizintechnik GmbH). SEPs recording are initiated in the emergency room or the angiosuit before the groin puncture and endovascular treatment, and continuous during the procedure. Because there may also be neurological damage during reperfusion (33), SEPs recordings are prolonged until patient leaves the angiography room and is transferred to the Acute Stroke Unit.

Both median nerves will be stimulated at wrist by means of surface adhesive electrodes. The investigators use supramaximal stimulation defined as the intensity that causes visually perceptible movement of the stimulated limb. The investigators apply square wave electrical pulses of 0.2 ms duration at a frequency of 5.7Hz. The investigators used a rate of 6.7 Hz if it is required according to the signal-to-noise ratio. SEPs are recorded in a referential fashion from the C3' (right median nerve stimulation) and C4' (left median nerve stimulation) positions and from a reference electrode at Fpz (international 10-20 system) or Cz' electrodes (2 cm behind Cz). The investigators use needle electrodes in conscious patients or "cork screw" electrodes in patients under general anesthesia during the thrombectomy procedure (Figure 1). The signal was digitally filtered (5-200 Hz bandpass) and analyzed within 80 msec time window poststimulus. Twenty to one hundred fifty trials were averaged depending on the signal-to-noise ratio.

The target signal is the presence of N20 response ipsilateral to the stroke site. Secondarily, the investigators also measure the amplitude and latency of N20 response both ipsilateral and contralateral to the stroke site. SEPs traces were analyzed at the moment of their recording by the examinators. Later, they also were analyzed by another blinded investigator to clinical outcome and SEPs monitoring.

Motor evoked potentials can not be performed because patients are awoke during the endovascular procedure according to the current standard of care

Primary Outcome The primary outcome is the functional independence at 7 days or discharge, defined by the modified Rankin scale score 0- 2. This early and more feasible outcome has a very high correlation with functional dependence at 90 days (Davalos A et al. Lancet Neurol 2017). Local certified assessors who are unaware of the SEPs monitoring findings evaluate the primary outcome variable in each patient by means of a structured interview.

Secondary outcomes Secondary clinical outcomes are the primary outcome evaluated at 90 days, the severity of disability at 7 days and 90 days, according to the distribution of scores on the modified Rankin scale (shift analysis), severe disability (score of 5) and death (score of 6) are combined into a single, worst category; early dramatic response to treatment (defined as a decrease in the NIHSS score of 8 or more points from baseline or an NIHSS score of 0 to 2 at 24 hours); and neurologic improvement at 24 hours defined as a decrease in the NIHSS score of 4 or more points from baseline).

Secondary neuroimaging variables are adjudicated infarct volume on CT or MRI at 24 hours; postprocedural revascularization classified as modified TICI scale 2b or 3 (indicating reperfusion of more than 50% of the affected territory); degree of vessel revascularization on CT angiography (CTA) or MR angiography (MRA) at 24 hours by using AOL scale or TCD by using TIMI score. In a subgroup of patients with pre- and post-MT multimodal MR or CTP, it will be calculated tissue perfusion recovery as the reperfusion index (TMax6s pre-MT x TMax6s post-MT)/TMax6s pre-MT). Lately, baseline imaging variables are also studied as potential predictors of recovery

Safety variables Safety outcomes are the rates of death and symptomatic intracranial hemorrhage at 90 days, as confirmed on neuroimaging (CT or MRI) evaluated by blinded investigators, according to the definition used in the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST). Evaluators also use the definition of symptomatic intracranial hemorrhage that was used in the second European-Australasian Acute Stroke Study (ECASS II) An independent investigator adjudicates procedure-related complications. Blood pressure variations during the procedure are also recorded.

Statistical Analysis All analyses will be performed in the total monitored patients (feasibility analysis). The primary measure of the effect size will be the unadjusted sensitivity and specificity (and their 95%CI) of the N20 response on SEPs prior to MT in predicting functional independence at 7 days or at discharge if earlier after treatment in patients with acute stroke and anterior large vessel occlusion.

According to our preliminary results, preestablished effect size is a true-positive rate of positive detection (functional independence) of > 92% (sensitivity) retaining a good rate of true-negative of negative detection (functional dependence) >90% (negative predictive value). In order to maintain the 95% low confidence intervals over 85% in both proportions, and considering a rate of negative detection of 28.6%, 228 patients are needed, 65 without N20 response and 163 with positive detection of N20 response. The adjusted predictive value of the N20 biomarker on functional independence after MT will be analyzed by binary logistic regression and its predictive value on the full range of disability (shift analysis) by ordinal logistic regression. The investigators will construct different regression models with other clinical predictors available at the prehospital setting and with those determined after hospital admission, including clinical and easy assessable imaging predictors. This analysis will give the independent predictive power of the N20 response for a potential treatment decision-making. The investigators will also evaluate the predictive binary effect of the N20 as a function of time from onset of symptoms to the first SEP stimulation and as a function of time from onset of symptoms to revascularization. Secondary analyses will include unadjusted association of N20 response with secondary clinical and neuroimaging outcomes and safety variables.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke with a demonstrated occlusion in the anterior circulation (M1 or M2 segment of middle cerebral artery with or without ipsilateral internal carotid artery (ICA)significant stenosis or occlusion diagnosed by CT angiography (CTA) or angio-MRI) undergoing urgent thrombectomy procedure.
* Prestroke functional independence of 2 or less on the modified Rankin scale (ranging from 0 [no symptoms] to 6 [death]),
* Baseline score of at least 6 points on the National Institutes of Health Stroke Scale (NIHSS), which ranges from 0 to 42, with higher values indicating more severe deficit.

Exclusion Criteria:

* Evidence by imaging of a large ischemic core, as indicated by an Alberta Stroke Program Early Computed Tomography Score (ASPECTS) of less than 5 on computed tomography (CT) without the use of contrast material or a score of less than 4 on diffusion-weighted magnetic resonance imaging (MRI) (ASPECTS values range from 0 to 10, with higher values indicating less infarct burden). These cutoff values of the ischemic core have been selected in agreement with the treatment effect showed in the HERMES trial meta-analysis collaboration (Presented at the International Stroke Conference, Houston, 2017).
* Well-documented history of neuromuscular disorders, stroke or central nervous system tumors that could interfere in the SEPs assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from our influence area (Barcelones-Nord-Maresme) ,other parts of Catalonia or people in this area at the moment of the acute stroke, arriving to our hospital because of an acute stroke of the anterior brain circulation, fulfilling criteria of endovascular urgent therapy
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Functional independence at 7 days or discharge | Baseline to 7 days or the day of discharge from hospital if it happens before the 7th day
  The primary outcome is the functional independence at 7 days or discharge, defined by the modified Rankin scale score 0- 2. This early and more feasible outcome has a very high correlation with functional dependence at 90 days (Davalos A et al. Lancet Neurol 2017). Local certified assessors who are unaware of the SEPs monitoring findings evaluate the primary outcome variable in each patient by means of a structured interview.

SECONDARY OUTCOMES:
Functional independence at 90 days from the stroke | Baseline to 90 days
  Secondary clinical outcomes are the primary outcome evaluated at 90 days, the severity of disability at at 7 days and 90 days, according to the distribution of scores on the modified Rankin scale (shift analysis), severe disability (score of 5) and death (score of 6) are combined into a single, worst category; early dramatic response to treatment (defined as a decrease in the NIHSS score of ≥8 from baseline or an NIHSS score of 0 to 2 at 24 hours); and neurologic improvement at 24 hours (defined as a decrease in the NIHSS score of ≥4 points from baseline).
Early dramatic response to treatment | Baseline to 24 hours
  decrease in the NIHSS score of 8 or more from baseline or an NIHSS score of 0 to 2 at 24 hours);
Neurologic improvement | Baseline to 24 hours
  Decrease in the NIHSS score of 4 or more points from baseline
Clinical status | Baseline to 7 days or the day of discharge from hospital if it happens before the 7th day
  NIHSS score at 24 hours and at 7 days or discharge from hospital if it happens before the 7th day
Infarct volume at 24 hours | Baseline to 24 hours
  Infarct volume on CT or MRI at 24 hours
Postprocedural revascularization | Baseline to end of thrombectomy treatment, an average of 1 hour
  Degree of revascularization classified as modified TICI scale 2b or 3 (indicating reperfusion of more than 50% of the affected territory)
Vessel revascularization | Baseline to 24 hours
  Degree of vessel revascularization on CT angiography (CTA) or MR angiography (MRA) at 24 hours by using AO scale or TCD by using TIMI score
Perfusion recovery | Baseline to end of thrombectomy treatment, an average of 1 hour
  In a subgroup of patients with pre- and post-MT multimodal MR or CTP, we calculate tissue perfusion recovery as the reperfusion index (TMax6s pre-MT x TMax6s post-MT)/TMax6s pre-MT)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Dávalos Errando, PhD, Principal Investigator — Fundació Institut d'Investigació en Ciències de la Salut Germans Trias iPujol
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Saver JL, Goyal M, van der Lugt A, Menon BK, Majoie CB, Dippel DW, Campbell BC, Nogueira RG, Demchuk AM, Tomasello A, Cardona P, Devlin TG, Frei DF, du Mesnil de Rochemont R, Berkhemer OA, Jovin TG, Siddiqui AH, van Zwam WH, Davis SM, Castano C, Sapkota BL, Fransen PS, Molina C, van Oostenbrugge RJ, Chamorro A, Lingsma H, Silver FL, Donnan GA, Shuaib A, Brown S, Stouch B, Mitchell PJ, Davalos A, Roos YB, Hill MD; HERMES Collaborators. Time to Treatment With Endovascular Thrombectomy and Outcomes From Ischemic Stroke: A Meta-analysis. JAMA. 2016 Sep 27;316(12):1279-88. doi: 10.1001/jama.2016.13647. PMID 27673305
- [Background] Lopez-Cancio E, Jovin TG, Cobo E, Cerda N, Jimenez M, Gomis M, Hernandez-Perez M, Caceres C, Cardona P, Lara B, Renu A, Llull L, Boned S, Muchada M, Davalos A. Endovascular treatment improves cognition after stroke: A secondary analysis of REVASCAT trial. Neurology. 2017 Jan 17;88(3):245-251. doi: 10.1212/WNL.0000000000003517. Epub 2016 Dec 9. PMID 27940648
- [Background] Davalos A, Cobo E, Molina CA, Chamorro A, de Miquel MA, Roman LS, Serena J, Lopez-Cancio E, Ribo M, Millan M, Urra X, Cardona P, Tomasello A, Castano C, Blasco J, Aja L, Rubiera M, Gomis M, Renu A, Lara B, Marti-Fabregas J, Jankowitz B, Cerda N, Jovin TG; REVASCAT Trial Investigators. Safety and efficacy of thrombectomy in acute ischaemic stroke (REVASCAT): 1-year follow-up of a randomised open-label trial. Lancet Neurol. 2017 May;16(5):369-376. doi: 10.1016/S1474-4422(17)30047-9. Epub 2017 Mar 16. PMID 28318984
- [Result] Alicia Martinez-Piñeiro , Giuseppe Lucente, María Hernandez-Perez, Jordi Cortés, Andrea Arbex, Natalia Pérez de la Ossa, Alba Ramos-Fransí, Miriam Almendrote, Mònica Millán, Meritxell Gomis, Laura Dorado, Carlos Castaño, Sebastián Remollo, Patricia Cuadras, Alicia Garrido, Nicolau Guanyabens, Joaquim Broto, Elena López-Cancio, Jaume Coll-Canti, Antoni Dávalos and PROMISE (Somatosensory Evoked POtEntials MonItoring During Acute Ischemic StrokE) Study Group. Prognostic Accuracy of N20 Somatosensory Potential in Patients With Acute Ischemic Stroke and Endovascular Thrombectomy Stroke: Vascular and Interventional Neurology. 2023 | Volume 3, Issue 5: e000735, originally publishedJune 14, 2023, https://doi.org/10.1161/SVIN.122.000735